CLINICAL TRIAL: NCT04124614
Title: A Phase 3, Multicenter, Randomized, Double-blind Trial of Brexpiprazole as Combination Therapy With Sertraline in the Treatment of Adults With Post-traumatic Stress Disorder
Brief Title: Brexpiprazole as Combination Therapy With Sertraline in Treatment of Adults With PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 331-201-00071
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — brexpiprazole; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Other): All enrolled participants received brexpiprazole-matched placebo tablets and sertraline-matched placebo tablets during the 1-week placebo run-in period.
  Interventions: Other: Placebo
- Brexpiprazole + Sertraline (Experimental): Randomized participants received brexpiprazole as a flexible dose 2 milligrams (mg) to 3 mg, orally, once daily (QD) along with sertraline, at a fixed dose of 150 mg, orally, QD from Week 1 to Week 12 of the double-blind treatment (DBT) period.
  Interventions: Drug: Brexpiprazole; Drug: Sertraline
- Sertraline + Placebo (Experimental): Randomized participants received sertraline, 150 mg, orally, QD along with sertraline matching placebo, orally, QD from Week 1 to Week 12 of the DBT period.
  Interventions: Drug: Sertraline; Other: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — 3 mg pill
  Other Names: Rexulti
  Arms: Brexpiprazole + Sertraline
Drug: Sertraline — 150 mg pill
  Other Names: Zoloft
  Arms: Brexpiprazole + Sertraline; Sertraline + Placebo
Other: Placebo — Pill
  Arms: Placebo; Sertraline + Placebo

SUMMARY:
This will be a 12-week, multicenter, randomized, double-blind trial evaluating the efficacy, safety, and tolerability of brexpiprazole + sertraline combination treatment in adult participants with Post-Traumatic Stress Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 to 65 years of age, inclusive, at the time of informed consent.
* Participants who have PTSD, diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), and confirmed by the Mini International Neuropsychiatric Interview (MINI).
* Onset of symptoms meeting the DSM-5 criteria for PTSD symptoms for a minimum of 6 months prior to screening.

Exclusion Criteria:

* The index traumatic event that led to the develop of PTSD took place > 9 years before screening.
* The index traumatic event occurred before age 16.
* Participants who have experienced a traumatic event within 3 months of screening.
* Participants who are receiving disability payments because of PTSD or any other psychiatric disorder; unless the disability payments will not be impacted by potential improvements demonstrated in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Davis LL, Behl S, Lee D, Zeng H, Skubiak T, Weaver S, Hefting N, Larsen KG, Hobart M. Brexpiprazole and Sertraline Combination Treatment in Posttraumatic Stress Disorder: A Phase 3 Randomized Clinical Trial. JAMA Psychiatry. 2025 Mar 1;82(3):218-227. doi: 10.1001/jamapsychiatry.2024.3996. PMID 39693081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 450 participants took part in the study at 61 investigative sites in the United States from 17 October 2019 to 08 August 2023.
Pre-assignment Details: Participants with a diagnosis of post-traumatic stress disorder (PTSD) were first enrolled in a placebo run-in period. At the end of placebo run-in period, participants were randomized in a 1:1 ratio to receive either Brexpiprazole + Sertraline or Sertraline + Placebo in the double-blind treatment (DBT) period.
Groups:
- Brexpiprazole + Sertraline: Randomized participants received brexpiprazole as a flexible dose 2 milligrams (mg) to 3 mg, orally, once daily (QD) along with sertraline, at a fixed dose of 150 mg, orally, QD from Week 1 to Week 12 of the DBT period.
Period: Placebo Run-in Period
Arm/Group | Placebo | Brexpiprazole + Sertraline | Sertraline + Placebo
Started | 450 | 0 | 0
Completed | 416 | 0 | 0
Not Completed | 34 | 0 | 0
Not completed — Not Randomized | 34 | 0 | 0
Period: Double Blind Treatment Period
Arm/Group | Placebo | Brexpiprazole + Sertraline | Sertraline + Placebo
Started | 0 | 214 | 202
Randomized Sample (Randomized Sample included all participants randomized into this trial.) | 0 | 214 | 202
Enriched Randomized Sample (Enriched Randomized Sample included all participants, randomized satisfying Enriched Participants Criteria, where Enriched Participants Criteria: Clinician-Administered PTSD Scale for Diagnostic & Statistical Manual of Mental Disorders,5th edition [DSM-5] (CAPS-5) total score of at least 27 at randomization visit (Week 1), & an improvement (reduction in CAPS-5 total score) in CAPS-5 total score of less than 50% at end of placebo run-in phase (from baseline to randomization visit [Week 1]).) | 0 | 160 | 150
FAS Enriched Sample (FAS for Enriched Participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score.) | 0 | 149 | 137
Safety Sample (Safety Sample included all participants in the randomized sample who were administered at least one dose of double-blind investigational medicinal product (IMP).) | 0 | 205 | 196
Completed | 0 | 137 | 113
Not Completed | 0 | 77 | 89
Not completed — Adverse Event | 0 | 7 | 22
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 18 | 25
Not completed — Non-Compliance With Study Drug | 0 | 5 | 5
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Protocol Deviation | 0 | 10 | 4
Not completed — Withdrawal by Subject | 0 | 26 | 22
Not completed — Reason Not Specified | 0 | 11 | 7

BASELINE CHARACTERISTICS:
Population: Randomized Sample included all participants randomized into this trial (DBT period).
Groups:
- Brexpiprazole + Sertraline: Randomized participants received brexpiprazole as a flexible dose 2 mg to 3 mg, orally, QD along with sertraline, at a fixed dose of 150 mg, orally, QD from Week 1 to Week 12 of the DBT period.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole + Sertraline | Sertraline + Placebo | Total
Number analyzed (Participants) | 214 | 202 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.7) | 36.8 (12.1) | 37.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 152 | 310
  Male | 56 | 50 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 147 | 144 | 291
  Black or African American | 50 | 38 | 88
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 4 | 9 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 32 | 61
  Not Hispanic or Latino | 183 | 167 | 350
  Unknown | 0 | 1 | 1
  Other | 2 | 2 | 4
CAPS-5 Total Severity Score [Mean (Standard Deviation); unit: score on a scale] — CAPS-5=structured interview designed to assess PTSD diagnostic status & symptoms severity as defined by DSM-5. CAPS-5 total score was calculated by summing severity scores for 20 DSM-5 PTSD symptoms (items 1-20) from following categories: Category B: Intrusion symptoms (5 items); Category C: Avoidance symptoms (2 items); Category D: Cognition & mood symptoms (7 items); Category E: Arousal & reactivity symptoms (6 items). Each symptom was scored 0=Absent to 4=Extreme/incapacitating, yielding a score range of 0-80. Higher scores indicate worse outcome. Population: FAS for Enriched participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score.
  score on a scale
    number analyzed (Participants) | 149 | 137 | 286
    (all) | 38.3 (7.2) | 38.8 (8.0) | 38.6 (7.6)
Clinical Global Impression - Severity (CGI-S) Score [Mean (Standard Deviation); unit: score on a scale] — CGI-S=standardized clinician-administered global rating scale measuring disease severity. To assess CGI-S, rater/investigator answered following question:"Considering your total clinical experience with this particular population,how mentally ill is participant at this time?"Response choices include:0=not assessed; 1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; & 7=among most extremely ill participants. Score 0 (not assessed) was to be set to missing. CGI-S is a 7-point scale from 1-7. Higher score =higher disease severity. Population: FAS for Enriched participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score. Number of participants analyzed is the number of participants with data available for CGI-S score at the Baseline.
  score on a scale
    number analyzed (Participants) | 148 | 137 | 285
    (all) | 4.6 (0.6) | 4.6 (0.6) | 4.6 (0.6)
Brief Inventory of Psychosocial Functions (B-IPF) Score [Mean (Standard Deviation); unit: score on a scale] — The B-IPF is a short patient-reported questionnaire consisting of 7 questions which measure PTSD-specific psychosocial function on a 7-point Likert scale (0 = not at all to 6 = very much, and a not applicable option) with a recall period of 30 days. It measures the concepts of romantic relationships, parenting, family, friendships and socializing, work, education, and self-care. Total score ranges from 0-100 and is calculated by summing the completed scale items, dividing by the maximum possible score of all items and multiplying by 100. Higher scores indicate greater impairment. Population: FAS for Enriched participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score. Number of participants analyzed is the number of participants with data available for B-IPF score at the Baseline.
  score on a scale
    number analyzed (Participants) | 142 | 129 | 271
    (all) | 65.2 (21.1) | 64.3 (22.9) | 64.8 (21.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score
Description: CAPS-5 is a structured interview designed to assess PTSD diagnostic status & symptoms severity as defined by DSM-5. CAPS-5 total score was calculated by summing severity scores for 20 DSM-5 PTSD symptoms (items 1-20) from following categories: Category B: Intrusion symptoms (5 items); Category C: Avoidance symptoms (2 items); Category D: Cognition & mood symptoms (7 items); Category E: Arousal & reactivity symptoms (6 items). CAPS-5 total score was imputed by adding all subscores from categories B, C, D, E. Each symptom was scored 0= Absent to 4= Extreme/incapacitating, yielding a score range of 0-80. Higher scores indicate worse outcome. Least squares (LS) mean was determined by Mixed-effect model repeated measures (MMRM) method with fixed class effect terms for treatment, trial site, visit, previous treatment intervention for PTSD (Yes/No), & an interaction term of treatment by visit, & include the interaction term of baseline values of CAPS-5 total score by visit as a covariate.
Time Frame: Baseline (Week 1), Week 10
Population: FAS for Enriched participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole + Sertraline | Sertraline + Placebo
Number analyzed (Participants) | 148 | 134
score on a scale | -19.19 (1.17) | -13.61 (1.24)
Statistical Analysis 1: Comparison: Brexpiprazole + Sertraline vs Sertraline + Placebo; Test type: Superiority — MMRM method with model terms: treatment, (pooled) study center, previous pharmacological treatment intervention for PTSD (yes/no), visit, treatment by visit and baseline by visit interaction; p = 0.0007, MMRM; Treatment Difference = -5.59, 95% CI 2-sided [-8.79 to -2.38]

2. Secondary Outcome: Change in Clinical Global Impression - Severity (CGI-S) Score
Description: The CGI-S is a standardized, clinician-administered global rating scale that measures disease severity. To assess it, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices include: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. The score 0 (not assessed) was be set to missing. The CGI-S is therefore a 7-point scale from 1 through 7. A higher score on the CGI-S represents a higher severity of disease. LS mean was determined by MMRM method with fixed class effect terms for treatment, trial site, visit, previous treatment intervention for PTSD (Yes/No), & an interaction term of treatment by visit, & include the interaction term of baseline values of CAPS-5 total score by visit as a covariate.
Time Frame: Baseline (Week 1), Week 10
Population: FAS for Enriched participants included those participants in the Enriched Randomized Sample who received at least 1 dose of double-blind IMP, had a baseline value (Week 1) and at least 1 post baseline efficacy evaluation for CAPS-5 total score. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole + Sertraline | Sertraline + Placebo
Number analyzed (Participants) | 148 | 137
score on a scale | -1.54 (0.10) | -1.08 (0.11)
Statistical Analysis 1: Comparison: Brexpiprazole + Sertraline vs Sertraline + Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0019, MMRM; Treatment Difference = -0.47, 95% CI 2-sided [-0.76 to -0.17]

3. Secondary Outcome: Change in Brief Inventory or Psychosocial Functions (B-IPF) Score
Description: The B-IPF is a short patient-reported questionnaire consisting of 7 questions which measure PTSD-specific psychosocial function on a 7-point Likert scale (0 = not at all to 6 = very much, and a not applicable option) with a recall period of 30 days. It measures the concepts of romantic relationships, parenting, family, friendships and socializing, work, education, and self-care. Total score ranges from 0-100 and is calculated by summing the completed scale items, dividing by the maximum possible score of all items and multiplying by 100. Higher scores indicate greater impairment. LS mean was determined by MMRM method with fixed class effect terms for treatment, trial site, visit, previous treatment intervention for PTSD (Yes/No), & an interaction term of treatment by visit, & include the interaction term of baseline values of CAPS-5 total score by visit as a covariate.
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexpiprazole + Sertraline | Sertraline + Placebo
Number analyzed (Participants) | 104 | 97
score on a scale | -33.80 (2.84) | -21.77 (2.97)
Statistical Analysis 1: Comparison: Brexpiprazole + Sertraline vs Sertraline + Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0016, MMRM; Treatment Difference = -12.03, 95% CI 2-sided [-19.44 to -4.62]

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to 21 days after the last dose (Up to Week 15)
Description: Safety Sample included all participants in the randomized sample who were administered at least one dose of double-blind IMP.
Arm/Group | Brexpiprazole + Sertraline | Sertraline + Placebo
All-Cause Mortality (participants affected / at risk) | 0/205 | 1/196
Serious Adverse Events (participants affected / at risk) | 1/205 | 4/196
Other Adverse Events (participants affected / at risk) | 68/205 | 58/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + Sertraline (N=205) | Sertraline + Placebo (N=196)
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + Sertraline (N=205) | Sertraline + Placebo (N=196)
Diarrhoea (Gastrointestinal disorders) | 9 | 13
Nausea (Gastrointestinal disorders) | 25 | 23
Fatigue (General disorders) | 14 | 8
Weight Increased (Investigations) | 12 | 3
Headache (Nervous system disorders) | 10 | 17
Somnolence (Nervous system disorders) | 11 | 5
Tremor (Nervous system disorders) | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04124614/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04124614/SAP_001.pdf